CLINICAL TRIAL: NCT00135655
Title: A Randomized, Double-Masked, Parallel, Group, Multi-Center, Dose Ranging Pilot Study of Denufosol Tetrasodium (INS37217) Intravitreal Injection in Subjects With Post Cataract Extraction Macular Edema
Brief Title: A Study of Denufosol Tetrasodium Intravitreal Injection in Subjects With Post Cataract Extraction Macular Edema
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-104
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Macular Edema, Cystoid
Keywords: macular edema; post cataract extraction; cystoid macular edema; post cataract extraction macular edema
MeSH Terms: conditions — Macular Edema | interventions — denufosol tetrasodium; Intravitreal Injections

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217) Intravitreal Injection

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of three dose strengths of the study drug in subjects with post cataract extraction macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Have persistent post cataract extraction macular edema whose condition is stable
* Have no change in medication regimen of immunosuppressive or anti-inflammatory agents; steroidal or non-steroidal agents for a specified period of time prior to randomization
* Have at least one eligible eye to be treated in the study
* Have an optical coherence tomography (OCT) scan with a qualifying retinal thickness in the study eye
* Have macular edema confirmed by fluorescein angiography

Exclusion Criteria:

* Have proliferative vitreoretinopathy greater than grade B in either eye
* Have ocular disorders in the study eye that may confound interpretation of study results
* Have ophthalmic disorders in the study eye that may influence final visual acuity and/or fluorescein angiography interpretation
* Have had cataract surgery in the study eye in the past 2 months, YAG laser capsulotomy within the past 1 month, or any other intraocular surgery within the past 90 days
* Have uncontrollable elevated intraocular pressure (IOP) or advanced glaucoma
* Have had any periocular or intravitreal injection of corticosteroids in the study eye within 3 months
* Have had any ocular implant device for the delivery of therapeutic agents
* Be taking any excluded medications that could obscure or confound study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08

PRIMARY OUTCOMES:
safety
tolerability
retinal thickness
visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director — Merck Sharp & Dohme LLC